CLINICAL TRIAL: NCT03483805
Title: Randomized, Double-blind, Controlled and Parallel Study of the Effect of a New Nutritional Solution to Improve Intestinal Permeability in Celiac Patients
Brief Title: Effects of a Nutritional Solution to Improve Intestinal Permeability in Celiac Patients
Acronym: Protalsafe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Guaranteed Gluten Free (GGF) (Industry)
Collaborators: Institut Polytechnique UniLaSalle (Unknown); Institut Pasteur de Lille (Other); Association Française des Intolérants au Gluten (AFDIAG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-A00330-51
Record Dates: First submitted 2018-03-19; First posted 2018-03-30 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Celiac Disease
Keywords: synbiotic; nutrition; permeability; gluten free diet; quality of life; digestive comfort
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Protalsafe product, daily, 12 weeks
  Interventions: Dietary Supplement: Protalsafe
- Placebo (Placebo Comparator): Placebo product, daily, 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Protalsafe — mix of prebiotic, probiotic and plant extract in powder form, to be diluted in water
  Arms: Treatment
Dietary Supplement: Placebo — maize maltodextrin in powder form, to be diluted in water
  Arms: Placebo

SUMMARY:
Celiac disease (or gluten intolerance) is recognized as one of the most common chronic diseases: prevalence of 1 in 100 to 1/300 people in Europe and the United States. To date, the treatment consists of a total elimination of any source of gluten from the diet. This eviction generates many daily constraints that would explain that more than 50% of patients do not follow this diet correctly. Hidden sources of gluten in a number of foods also carry the burden of this difficulty in effective exclusion. The objective of the ProtAlSafe study is to develop an innovative nutritional approach in the form of a dietary supplement to improve quality of life of patients. The product is not intended to replace a strict gluten-free diet but to propose a nutritional approach in the form of a dietary supplement to improve quality of life of patients. The expected benefits for people consuming the test product are an overall improvement in quality of life and an improvement in biological markers (intestinal permeability, chronic inflammation, etc.) associated with celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* celiac disease diagnosis at least 1 year ago
* diagnosis proven through biopsy report or general practioner letter or health insurance cover
* not following a strict gluten free diet (Pavie score 1-3)
* covered by health insurance
* not in exclusion period from another study

Exclusion Criteria:

* pregnant, breastfeeding women or planing pregnancy
* gluten intolerance of non celiac origin or any other dietary intolerance of allergy
* digestive pathology other than celiac disease
* chronic transit problems (diarrhoea or constipation)
* uncontrolled pathology
* diabetes
* medical treatment impacting outcome markers (corticosteroids, NSAIDS, immune suppressor drugs, pancreatic enzymes, amphetamines)
* recent or regular intake of prebiotics, probiotics, food supplements including B vitamins, iron or calcium.
* antibiotics in the past month
* excessive alcohol intake
* drug user
* planing to change tobacco use
* any other reason why the investigator feels the subject may not be compliant
* adults under judicial protection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Lactulose/mannitol recovery in 5-hour urine sample | after 12 weeks of treatment
  ratio of the two sugars following ingestion
serum zonulin | after 12 weeks of treatment
  circulating concentration

SECONDARY OUTCOMES:
microbiota profile | baseline and after 12 weeks of treatment
  taxonomic sequencing
digestive health | baseline and after 12 weeks of treatment
  gastrointestinal symptoms rating scale (GSRS), 13 questions with answers rating from 0 to 3
digestive comfort | baseline and after 12 weeks of treatment
  visual analogic scale on digestive symptoms, 5 questions with 10cm scale rating from no symptoms (left) to worsening
quality of life- digestive health | baseline and after 12 weeks of treatment
  celiac disease quality of life questionnaire (F-CDQ), subset of digestive questions
quality of life | baseline and after 12 weeks of treatment
  celiac disease quality of life questionnaire (F-CDQ)
circulating inflammation markers | baseline and after 12 weeks of treatment
  concentration of cytokines interleukin-6, tumor necrosis factor-alpha and interleukin-10

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Pasteur de Lille, Lille, France